CLINICAL TRIAL: NCT06759506
Title: Can Perfusion Index and Cerebral Oxygen Saturation Trends Predict Low Cardiac Output in Pediatric Cardiovascular Surgeries
Status: Not yet recruiting | Type: Observational
Sponsor: Bozyaka Training and Research Hospital (Other)
Collaborators: Basaksehir Cam & Sakura City Hospital (Unknown)
Responsible Party: Principal Investigator, Ezgi Direnç YÜCEL, Consultant Anaesthetist, Bozyaka Training and Research Hospital
Other Study IDs: ZeynepTez
Record Dates: First submitted 2024-12-28; First posted 2025-01-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Perfusion Index and Cerebral NIRS Trends in Low Cardiac Output Syndrome
Keywords: Congenital Cardiac Surgery; Perfusion Index; Low Cardiac Output Syndrome
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
In this prospective, observational study, we aim to investigate whether routinely monitored Perfusion Index (PI) and cerebral oxygen saturation (NIRS) values in pediatric patients aged 0-6 undergoing congenital heart surgery are associated with Low Cardiac Output Syndrome. Pediatric patients aged 0-6 years undergoing congenital heart surgery will be followed primarily for Cerebral Near-Infrared Reflectance Spectroscopy, and Perfusion Index (PI) values both in the operating room during the operation, and in the Pediatric Cardiac Intensive Care Unit during the first 24 hours postoperatively. The patients with Low Cardiac Output Syndrome will be recorded, and the changes in Cerebral Near-Infrared Reflectance Spectroscopy, and Perfusion Index (PI) values will be evaluated to determine whether they can predict low cardiac output.

DETAILED DESCRIPTION:
All patients will have their demographic characteristics routinely recorded, including preoperative echocardiographic measurements and initial hemodynamic monitoring parameters before surgery. Operative details such as operation and anesthesia durations, bypass and cross-clamp times, heart rate, blood pressure, NIRS values, urine output, blood gas parameters, and use of inotropes and blood products will also be documented.

During the first 24 hours postoperatively, at 0, 6, 12, and 24 hours, bedside visits will be conducted to record the following parameters per patient: heart rate, blood pressure, urine output, peripheral and central body temperature, capillary refill time, inotropic requirement, blood product requirement, serum lactate level, central venous oxygen saturation, cerebral Near-Infrared Reflectance Spectroscopy, and Perfusion Index (PI) values.

Preoperative and perioperative parameters will be recorded by anesthesia technicians and anesthesiologists; postoperative parameters will be recorded by Pediatric Cardiac Intensive Care physicians and nurses. The monitoring methods and parameters followed in the research are routine in pediatric cardiac surgery during intraoperative and postoperative periods.

Echocardiographic findings immediately post-operation and within the first 24 hours will be noted to observe the presence and severity of Low Cardiac Output Syndrome.

With these recorded parameters, the presence of Low Cardiac Output Syndrome within the first 24 hours postoperatively will be examined, alongside the assessment of inotropic requirement, need for dialysis, use of extracorporeal membrane oxygenation, revision surgeries, mortality, and morbidity. This data will be used to investigate the frequency of Low Cardiac Output Syndrome, its causes, and the relationship with NIRS and PI in pediatric patients aged 0-6 undergoing congenital cardiac surgery.

The monitoring methods and parameters followed in the research are routine in pediatric cardiac surgery during intraoperative and postoperative periods. They do not require additional costs or manpower. The researchers will conduct the study in accordance with the Helsinki Declaration and Good Clinical Practice principles.

Every patient, whether enrolled in any study or not, will be routinely monitored by our team during anesthesia administration and post-anesthesia care (this monitoring practice includes regular visits, examinations, and follow-ups of our clinic's patients). Consent will be obtained from our patients for these practices, and no additional laboratory tests will be conducted for this study. Patients will receive their routine treatments as needed without any alterations. In this study, intraoperative and postoperative monitoring data that have been observed will be used.

Since no additional interventions beyond our routine practices will be undertaken, no circumstances threatening patient safety, problems, or complications are expected to arise At the conclusion of the study, all data will be entered into a computer and analyzed using the SPSS software. Statistical methods including chi-square test, student's t-test, and Mann-Whitney U test will be used for intergroup comparisons, with a significance level set at P ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0-6 years who undergo congenital heart surgery and develop low cardiac output syndrome

Exclusion Criteria:

* Patients older than 6 years
* Premature infants
* Patients who were operated on at external institutions and later transferred to our facility
* Patients with low cardiac output syndrome not related to the postoperative period

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 0-6 years who undergo congenital heart surgery and develop low cardiac output syndrome
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
PI in low cardiac output | 24 hours postoperatively
  Perfusion Index (PI) trends in pediatric cardiac surgery cases with low cardiac output
Serebral NIRS in low cardiac output | Intraoperatively and first 24 hours postoperatively
  Serebral NIRS in trends in pediatric cardiac surgery cases with low cardiac output

SECONDARY OUTCOMES:
Inotropic requirements | Intraoperatively and first 24 hours postoperatively
  Inotropic requirements in pediatric cardiac surgery cases with low cardiac output
Need for dialysis | 24 hours postoperatively
  Need for dialysis in pediatric cardiac surgery cases with low cardiac output
Need for ECMO (extracorporeal membrane oxygenation) | 24 hours postoperatively
  Need for ECMO in pediatric cardiac surgery cases with low cardiac output
Need for reoperation | 24 hours postoperatively
  Need for reoperation in pediatric cardiac surgery cases with low cardiac output
Mortality | 24 hours postoperatively
  Mortality in pediatric cardiac surgery cases with low cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: Funda Gümüş Özcan, Study Director — Istanbul Cam and Sakura City Hospital

IPD SHARING:
Plan to Share IPD: No